CLINICAL TRIAL: NCT04312334
Title: Improving the Supertowel: An Alternative Hand Cleaning Product for Emergencies
Acronym: Supertowel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Kelkar Education Trust's Scientific Research Centre, Mumbai (India) (Other); Real Relief Health ApS,Essen 26, 6000 Kolding, Denmark (Unknown); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: LSHTM ethics ref: 18006
Record Dates: First submitted 2020-03-12; First posted 2020-03-18 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-03

CONDITIONS: Escherichia Coli Change
Keywords: Escherichia Coli change; Hand-washing; Emergency settings; Hand-cleaning; Hygiene
MeSH Terms: interventions — Hand Disinfection; Soaps; Therapeutics

STUDY DESIGN:
Intervention Model Description: To test the efficacy of the Supertowel under the different conditions, we will use a crossover controlled study based and adapted on the protocol of the European Committee for Standardization (EN 1499) which is designed to evaluate the ability of hand-wash agents to eliminate transient pathogens from volunteers' hands without regard to resident microorganisms. This procedure is based on the "post-contamination treatment" of hands and involves the placement of the test organism (E. coli [ATCC 11229]) on the hands of test subjects, followed by exposure of the test product.The study will be organized in two rounds of tests.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be masked to treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Treatment 1 (Experimental): Treatment 1: Hand cleaning with the Supertowel for 15 seconds. The Supertowel will be soaked in water by submersing it completely in a bucket filled with tap water. The amount of water absorbed by the ST will be recorded by means of weighing the towel before and after soaking. The volunteers will use the soaked Supertowel for 15 seconds to clean their pre-contaminated hands.
  Interventions: Other: Treatment
- Treatment 2 (Experimental): Treatment 2: Hand cleaning with a Supertowel that is damp for 60 seconds The Supertowel will be soaked in water by submersing it completely in a bucket filled with tap water. The water on the Supertowel will then be squeezed out so that it is not dripping. The Supertowel will be weighed before soaking and after squeezing. Volunteers will clean their pre-contaminated hands with the damp Supertowel for 60 seconds.
  Interventions: Other: Treatment
- Treatment 3 (Experimental): Treatment 3: Hand cleaning for 60 seconds with a Supertowel that has been soaked in contaminated water.
  A Supertowel will be soaked in water which has artificially contaminated with non-pathogenic E.coli. The water will be designed to mimic highly contaminated grey water so it will be contaminated at 2,000 cfu/100 ml which is double the acceptable level of contamination for handwashing. Volunteers will clean their pre-contaminated hands with the contaminated Supertowel for 60 seconds.
  Interventions: Other: Treatment
- Treatment 4 (Experimental): Treatment 4: Hand cleaning for 60 seconds with a Supertowel that is visibly dirty and oily.
  The Supertowel will be made visibly dirty and oily for example, by immersing it in a mix of 10 grams of sterile soil (previously autoclaved), 1 ml of clean cooking oil and 100 ml of water .The Supertowel will be rubbed against itself to ensure the soil and oil are spread out across the surface of the Supertowel. Volunteers will clean their pre-contaminated hands with the dirty Supertowel for 60 seconds.
  Interventions: Other: Treatment
- Treatment 5 (Experimental): Treatment 5: Hand cleaning for 30 seconds with a Supertowel that is visibly dirty and oily and it is soaked in whater which has artificially contaminated with non-pathogenic E.coli.
  The Supertowel will be made visibly dirty and oily for example, by immersing it in a mix of 10 grams of sterile soil (previously autoclaved), 1 ml of clean cooking oil and 100 ml of water (which will be contaminated with E.coli).The Supertowel will be rubbed against itself to ensure the soil and oil are spread out across the surface of the Supertowel. Volunteers will clean their pre-contaminated hands with the dirty Supertowel for 30 seconds.
  Interventions: Other: Treatment
- Treatment 6 (Experimental): Treatment 6: Hand cleaning with the Supertowel which is fully dry for 60 seconds.
  Interventions: Other: Treatment
- Control 1 (Other): Control 1: Hand washing with bar soap and water for 15 seconds. The control group will wash their pre-contaminated hands with normal bar soap and water for 15 seconds. Hands from volunteers washed with soap will be allowed to dry for 3 minutes.
  Interventions: Other: Control
- Control 2 (Other): Control 2: Handwashing with bar soap and water for 60 seconds The control group will wash their pre-contaminated hands with normal bar soap and water for 60 seconds by following the "WHO guidelines for handwashing when hands are visibly soiled" (a diagram of the steps was given to them, appendix). After handwashing, hands will be allowed to dry for 3 minutes
  Interventions: Other: Control
- Control 3 (Other): Control 3: Handwashing with bar soap and contaminated water for 60 seconds. Water which is contaminated with non-pathogenic E.coli. at 2,000 cfu/100ml will be stored in a bucket which has a tap at the base. The control group volunteers will wash their hands with the contaminated water and bar soap for 60 seconds. They will follow the "WHO guidelines for handwashing when hands are visibly soiled" (a diagram of the steps will be given to them). After handwashing, hands will be allowed to dry for 3 minutes.
  Interventions: Other: Control
- Control 4 (Other): Control 4: Hand cleaning for 60 seconds with a clean Supertowel. The Supertowel will be soaked in water by submersing it completely in a bucket filled with tap water. The amount of water absorbed by the ST will be recordedby means of weighing the Supertowel before and after soaking. The control group will clean their pre-contaminated hands of with thesoaked Supertowel for 60 seconds.
  Interventions: Other: Treatment
- Control 5 (Other): Hand washing with bar soap and water for 30 seconds. The control group will wash their pre-contaminated hands with normal bar soap and water for 30 seconds. Hands from volunteers washed with soap will be allowed to dry for 3 minutes.
  Interventions: Other: Control

INTERVENTIONS:
Other: Control — Soap: Non-antimicrobial bar soap will be used as a reference product for four of the the experiments. Hand-cleaning with SuperTowel will be the reference produce for two of the experiments.
  Other Names: Hand-cleaning with Supertowel or hand-washing with soap
  Arms: Control 1; Control 2; Control 3; Control 5
Other: Treatment — The Supertowel is a durable fabric with a permanent anti-microbial treatment. The treated fabric must be dipped in water and then rubbed against the hands so that pathogens will be transferred to the fabric where they will be killed.
  Other Names: Treatment with SupeTowel
  Arms: Control 4; Treatment 1; Treatment 2; Treatment 3; Treatment 4; Treatment 5; Treatment 6

SUMMARY:
The Supertowel is a microfiber towel treated with a permanent anti-microbial bonding and has been designed as a soap alternative in emergency situations.The treated fabric must be dipped in water and then rubbed against the hands so that pathogens will be transferred to the fabric where they will be killed. Over the last two years the investigators have been able to prove, under controlled laboratory conditions, that hand cleaning with the Supertowel is more efficacious than handwashing soap and water. Another field study conducted by the investigators in a refugee camp in Northern Ethiopia indicated that the Supertowel is an acceptable and desirable product among crisis-affected populations and is likely to result in more frequent handwashing in these difficult circumstances.

The aim of this study is to develop greater evidence on whether the Supertowel remains is as efficacious when used under conditions which mimic "real-world hand cleaning conditions". This will be tested through a set of controlled laboratory experiments with healthy volunteers in India.

DETAILED DESCRIPTION:
The Supertowel is a microfiber towel treated with a permanent anti-microbial bonding and has been designed as a soap alternative in emergency situations.

The treated fabric must be dipped in water and then rubbed against the hands so that pathogens will be transferred to the fabric where they will be killed. Several laboratory test have demonstrated the bactericidal effect of the fabric against different bacteria. The Supertowel will kill microbes efficiently and within seconds once the microbe is on the towel. The Supertowel provides an alternative to large-scale soap distribution. It could be beneficial to emergency responders as it will be easier (smaller and lighter) to distribute and last longer than soap, negating the need for frequent distributions. The Supertowel will reduce water wastage associated with hand washing and reduce drainage problems that are often seen around hand washing facilities. The Supertowel will also be beneficial to those effected by emergencies as it can easily be carried by users all the time, making hand cleaning more convenient.

Over the last two years the investigators have been able to prove, under controlled laboratory conditions, that hand cleaning with the Supertowel is more efficacious than handwashing soap and water. Another field study conducted by the investigators in a refugee camp in Northern Ethiopia indicated that the Supertowel is an acceptable and desirable product among crisis-affected populations and is likely to result in more frequent handwashing in these difficult circumstances.

The aim of this study is to develop greater evidence on whether the Supertowel remains is as efficacious when used under conditions which mimic "real-world hand cleaning conditions". This will be tested through a set of controlled laboratory experiments with healthy volunteers in India. We will be testing the efficacy of the Supertowel as a hand-cleaning product using simulations of 'real-world' hand cleaning conditions.

To test the efficacy of the Supertowel under the different conditions, we will use a crossover controlled study based and adapted on the protocol of the European Committee for Standardization (EN 1499) which is designed to evaluate the ability of hand-wash agents to eliminate transient pathogens from volunteers' hands without regard to resident microorganisms. This procedure is based on the "post-contamination treatment" of hands and involves the placement of the test organism (E. coli [ATCC 11229]) on the hands of test subjects, followed by exposure of the test product.

The study will be organized in two rounds of tests. 32 healthy volunteers will be selected for the study. 16 volunteers will be invited for the first round and 16 more for the second round. Each volunteer will receive treatment with all the different procedures the same day of visit to the laboratory.

This is a single centre study conducted in KET's Scientific Research Centre, Mumbai (India). The recruitment and performance of tests will be done at KET's Scientific Research Centre, Mumbai (India) Laboratory of India.

ELIGIBILITY:
Inclusion Criteria:

To be eligible volunteers must:

* Be male and older than 18 years old.
* Be physically examined to ensure they are healthy and with healthy skin (without skin disorders like eczema, paronychia, scabies, abrasions, lacerations or skin allergy).
* Have short fingernails with no artificial nails.
* Have no history of drug allergy.
* Nothave taken any systemic antibiotic in the two weeks prior to the study, which could otherwise impair the efficacy of the product being tested.
* Remove all forms of jewellery from their hands prior to hand washing, since it has the potential of retain some bacteria, which could affect the recovery pre and post values of the test.

Exclusion Criteria:

* Unhealthy volunteers and volunteers with unhealthy skin, history of drug allergy, taken systemic antibiotics in the previous two weeks of the study will be excluded from the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Change of E.coli | 24 hours
  Reduction of bacteria (E.coli (ATCC 11229)) in pre-contaminated hands of volunteers after using the different test conditions. This procedure is based on the "post-contamination" treatment of hands and involves the placement of the test organism (E.coli (ATCC 11229)) on the hands of test subjects, followed by exposure of the test product. For both the Supertowel product or soap treatments, log10 counts from left and right hands of each subject were averaged separately, for both pre- and post-values. The arithmetic means of all individuals log10 changes values will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Belen Torondel, Dr, Principal Investigator — Dr
Locations (1):
- KETs Scientific Research Centre, Mumbai, India

IPD SHARING:
Plan to Share IPD: Yes
Once we have the results analyzed and published we are happy to share the results with other interested researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 years
Access Criteria: The PI and Co-Is will decide whether to grant release of the data based on these requests. Our intended policy will be to make data available to researchers, within 2 years of completion of the study. This is to make maximum use of data collected using public funding while protecting the intellectual property rights of the study team.

REFERENCES:
- [Result] Torondel B, Khan R, Holm Larsen T, White S. Efficacy of the SuperTowel(R): An Alternative Hand-washing Product for Humanitarian Emergencies. Am J Trop Med Hyg. 2019 May;100(5):1278-1284. doi: 10.4269/ajtmh.18-0860. PMID 30860009
- [Result] White S, Petz JF, Desta K, Holm Larsen T. Could the Supertowel be used as an alternative hand cleaning product for emergencies? An acceptability and feasibility study in a refugee camp in Ethiopia. PLoS One. 2019 May 6;14(5):e0216237. doi: 10.1371/journal.pone.0216237. eCollection 2019. PMID 31059540
- Available data/document: Individual Participant Data Set — https://bmcmedicine.biomedcentral.com/articles/10.1186/s12916-015-0532-z — Our data will be suitable for sharing in anonymised form.Potential users will learn about the data on the websites of the collaborating institutes, and links to the relevant data repositories will be available on those websites.The link will contain information on how to apply to use the data. We aim to offer controlled access to study data. Potential users of the data will be invited to register and provide information on their aims and proposed analyses of the data. The PI and Co-Is will decide whether to grant release of the data based on these requests. Our intended policy will be to make data available to researchers, within 2 years of completion of the study. This is to make maximum use of data collected using public funding while protecting the intellectual property rights of the study team.Restrictions or delays to sharing, with planned actions to limit such restrictions We would like to retain exclusive use for 2 years

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT04312334/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT04312334/ICF_001.pdf